CLINICAL TRIAL: NCT04305717
Title: Remote Dielectric Sensing (ReDS) for a SAFE Discharge in Patients With Acutely Decompensated Heart Failure: The ReDS-SAFE HF Study
Brief Title: Use of ReDS Technology in Patients With Acute Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Donna Mancini, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 19-2678
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure; Lung Congestion
Keywords: Clinical trial; Lung congestion; Heart failure; Diuretics
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The ReDS-SAFE HF trial is a 2-arm randomized clinical trial, in which inpatients with ADHF will be randomized to:
  1. Standard of care strategy, with a discharge scheme based on current clinical practice, or
  2. ReDS-guided strategy, with a discharge scheme based on specific target value given by the device.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant masking: Patients will be blinded to the treatment groups. ReDS tests will be performed for all study patients, but due to the inherent characteristics of this design, only the treating physicians will be blinded in the "standard of care" arm.
  Outcome assessor masking: Two independent cardiologist will assess the outcomes blinded to the intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ReDS-guided strategy (Experimental): For patients in this arm, daily measurements from the device will be revealed to the treating physician. Discharge can be planned when the clinical stability is achieved and the ReDS value is ≤35%. In case of a ReDS value >35%, treating physicians will follow a predefined algorithm before discharge to improve the results of ReDS test.
  Interventions: Device: ReDS-guided strategy
- Standard of care strategy (No Intervention): The drugs dosage, especially diuretics, will be selected according to the presence of symptoms and signs of systemic congestion and according to current recommendations. All the daily ReDS measurements will be blinded to the treating physician.

INTERVENTIONS:
Device: ReDS-guided strategy — A discharge scheme based on specific target value given by the device
  Arms: ReDS-guided strategy

SUMMARY:
Background: Fluid overload, especially pulmonary congestion, is one of the main contributors into heart failure (HF) readmission risk and it is a clinical challenge for clinicians. The Remote dielectric sensing (ReDS) system is a novel electromagnetic energy-based technology that can accurately quantify changes in lung fluid concentration noninvasively. Previous non-randomized studies suggest that ReDS-guided management has the potential to reduce readmissions in HF patients recently discharged from the hospital.

Aims: To test whether a ReDS-guided strategy during HF admission is superior to the standard of care during a 1-month follow up.

Methods: The ReDS-SAFE HF trial is an investigator-initiated, single center, single blind, 2-arm randomized clinical trial, in which ~240 inpatients with acutely decompensated HF at Mount Sinai Hospital will be randomized to a) standard of care strategy, with a discharge scheme based on current clinical practice, or b) ReDS-guided strategy, with a discharge scheme based on specific target value given by the device on top of the current clinical practice. ReDS tests will be performed for all study patients, but results will be blinded for treating physicians in the "standard of care" arm. The primary outcome will be a composite of unplanned visit for HF that lead to the use of intravenous diuretics, hospitalization for worsening HF, or death from any cause at 30 days after discharge. Secondary outcomes including the components of the primary outcome alone, length of stay, quality of life, time-averaged proportional change in the natriuretic peptides plasma levels, and safety events as symptomatic hypotension, diselectrolytemias or worsening of renal function.

Conclusions: The ReDS-SAFE HF trial will help to clarify the efficacy of a ReDS-guided strategy during HF-admission to improve the short-term prognosis of patients after a HF admission.

DETAILED DESCRIPTION:
Heart failure (HF) is an increasing epidemic and a major public health priority, affecting more than 6 million patients in the United States of America (1). Specially, acutely decompensated HF (ADHF) is the most common cause of hospitalization in adults older than 65 years, and is associated with high rates of morbidity and mortality. Despite advances in pharmacological treatment and early follow-up programs in HF patients, readmission rates remain unacceptably high (2).

Fluid overload is a key feature in the pathophysiology of ADHF and residual congestion at the time of hospital discharge is one of the main contributors into readmission risk (3-5). Typically, fluid overload has been assessed through symptoms and signs, as well as other tools such as chest X-ray, plasma biomarkers, and echocardiography (6). However, these methods are subject to significant inter-observer variability and can be unreliable for various reasons. Furthermore, recent studies have shown that overt signs of clinical congestion correlate poorly with hemodynamic congestion assessed by invasive means. In recent years, invasive hemodynamic measurements to inform medical management of congestion facilitated by implantable pulmonary artery pressure sensors have been shown to reduce HF readmissions (7). Unfortunately, due to its invasive nature as well as reimbursement and insurance coverage issues, its widespread adoption has been limited.

Thus, the use of a non-invasive assessment of volume status to guide HF management and identify a state of "euvolemia" is an attractive tool, particularly during admission and early phase after discharge, which is a vulnerable period for recurrent congestion (8). The Remote dielectric sensing (ReDS) system is a novel electromagnetic energy-based technology that can accurately quantify changes in lung fluid concentration noninvasively (9). Though limited experience from non-randomized studies suggest that ReDS-guided management has the potential to reduce readmissions in ADHF patients recently discharged from the hospital (10, 11), nevertheless data to substantiate the employment of such as strategy is lacking. The study team hypothesizes that a ReDS-guided strategy to measure the percent of lung water volume as a surrogate of congestion during HF hospitalization will help to determine the appropriate timing of discharge and will accordingly be associated with a better short-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Currently hospitalized for a primary diagnosis of HF, including symptoms and signs of fluid overload, regardless of left ventricular ejection fraction (LVEF), and a NT-proBNP concentration of ≥ 400 pg/L or a BNP concentration of ≥ 100 pg/L

Exclusion Criteria:

* Patient characteristics excluded from approved use of ReDS system: height <155cm or >190cm, BMI <22 or >39
* Patients discharged on inotropes, or with a left ventricular assist device or cardiac transplantation
* Congenital heart malformations or intra-thoracic mass that would affect right-lung anatomy
* End stage renal disease on hemodialysis
* Life expectancy <12 months due to non-cardiac comorbidities
* Participating in another randomized study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | 30 days after discharge
  A composite of unplanned visit for ADHF that lead to the use of intravenous diuretics, hospitalization for worsening HF, or death from any cause at 30 days after discharge.

SECONDARY OUTCOMES:
Number of unplanned visits | 30 days after discharge
  Unplanned visits for worsening HF will be defined as visits to the emergency department or unscheduled visits to the HF unit as a result of signs and/or symptoms of worsening HF that required iv diuretic treatment or diuretic increase with a hospital stay of <24 h.
Number of unplanned hospitalizations | 30 days after discharge
  Hospitalization for worsening HF will be defined as a stay in hospital for >24 h mainly as a result of signs and/or symptoms of worsening HF.
Length of stay | average of 7 days
  Length of stay of index hospitalization
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 7 days after discharge
  QoL evaluated by the KCCQ test which is a 23-item, self-administered instrument. Full scale range from 0-100, with higher scores reflecting better health status
New York Heart Association functional class | 7 days after discharge
  New York Heart Association functional classification from Class 1 (no symptom or limitation to Class IV (severe symptoms or severe limitation).
Orthodema Scale | 7 days after discharge
  Signs of systemic congestion by Orthodema scale. Full scale from 0 to 4, with higher score indicating worse health outcomes.
Breathlessness Visual Analog Scale | 7 days after discharge
  Signs of resolution of the breathlessness by visual analog scale. Full scale from 0 to 10, with higher score indicating better health outcomes.
Change in NT-proBNP/BNP plasma levels | baseline and 7 days after discharge
  Time-averaged proportional change in the NT-proBNP/BNP plasma levels at 7 days after discharge as compared from baseline
Serum Potassium | 7 days after discharge
  Serum potassium level to assess dyskalemia
Change in Creatinine level | baseline and 7 days after discharge
  Change in creatinine from at 7 days after discharge as compared to baseline
Systolic arterial pressure | 7 days after discharge
  Systolic arterial pressure to assess hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Mancini, Principal Investigator — Icahn School of Medicine
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Kociol RD, McNulty SE, Hernandez AF, Lee KL, Redfield MM, Tracy RP, Braunwald E, O'Connor CM, Felker GM; NHLBI Heart Failure Network Steering Committee and Investigators. Markers of decongestion, dyspnea relief, and clinical outcomes among patients hospitalized with acute heart failure. Circ Heart Fail. 2013 Mar;6(2):240-5. doi: 10.1161/CIRCHEARTFAILURE.112.969246. Epub 2012 Dec 18. PMID 23250981
- [Background] Gheorghiade M, Follath F, Ponikowski P, Barsuk JH, Blair JE, Cleland JG, Dickstein K, Drazner MH, Fonarow GC, Jaarsma T, Jondeau G, Sendon JL, Mebazaa A, Metra M, Nieminen M, Pang PS, Seferovic P, Stevenson LW, van Veldhuisen DJ, Zannad F, Anker SD, Rhodes A, McMurray JJ, Filippatos G; European Society of Cardiology; European Society of Intensive Care Medicine. Assessing and grading congestion in acute heart failure: a scientific statement from the acute heart failure committee of the heart failure association of the European Society of Cardiology and endorsed by the European Society of Intensive Care Medicine. Eur J Heart Fail. 2010 May;12(5):423-33. doi: 10.1093/eurjhf/hfq045. Epub 2010 Mar 30. PMID 20354029
- [Background] Amir O, Rappaport D, Zafrir B, Abraham WT. A novel approach to monitoring pulmonary congestion in heart failure: initial animal and clinical experiences using remote dielectric sensing technology. Congest Heart Fail. 2013 May-Jun;19(3):149-55. doi: 10.1111/chf.12021. Epub 2013 Jan 25. PMID 23350643
- [Background] Gargani L, Pang PS, Frassi F, Miglioranza MH, Dini FL, Landi P, Picano E. Persistent pulmonary congestion before discharge predicts rehospitalization in heart failure: a lung ultrasound study. Cardiovasc Ultrasound. 2015 Sep 4;13:40. doi: 10.1186/s12947-015-0033-4. PMID 26337295
- [Background] Abraham WT, Adamson PB, Bourge RC, Aaron MF, Costanzo MR, Stevenson LW, Strickland W, Neelagaru S, Raval N, Krueger S, Weiner S, Shavelle D, Jeffries B, Yadav JS; CHAMPION Trial Study Group. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. Lancet. 2011 Feb 19;377(9766):658-66. doi: 10.1016/S0140-6736(11)60101-3. PMID 21315441
- [Background] Amir O, Ben-Gal T, Weinstein JM, Schliamser J, Burkhoff D, Abbo A, Abraham WT. Evaluation of remote dielectric sensing (ReDS) technology-guided therapy for decreasing heart failure re-hospitalizations. Int J Cardiol. 2017 Aug 1;240:279-284. doi: 10.1016/j.ijcard.2017.02.120. Epub 2017 Mar 3. PMID 28341372
- [Background] Goldgrab D, Balakumaran K, Kim MJ, Tabtabai SR. Updates in heart failure 30-day readmission prevention. Heart Fail Rev. 2019 Mar;24(2):177-187. doi: 10.1007/s10741-018-9754-4. PMID 30488242
- [Background] Lala A, McNulty SE, Mentz RJ, Dunlay SM, Vader JM, AbouEzzeddine OF, DeVore AD, Khazanie P, Redfield MM, Goldsmith SR, Bart BA, Anstrom KJ, Felker GM, Hernandez AF, Stevenson LW. Relief and Recurrence of Congestion During and After Hospitalization for Acute Heart Failure: Insights From Diuretic Optimization Strategy Evaluation in Acute Decompensated Heart Failure (DOSE-AHF) and Cardiorenal Rescue Study in Acute Decompensated Heart Failure (CARESS-HF). Circ Heart Fail. 2015 Jul;8(4):741-8. doi: 10.1161/CIRCHEARTFAILURE.114.001957. Epub 2015 Jun 3. PMID 26041600
- [Background] Picano E, Gargani L, Gheorghiade M. Why, when, and how to assess pulmonary congestion in heart failure: pathophysiological, clinical, and methodological implications. Heart Fail Rev. 2010 Jan;15(1):63-72. doi: 10.1007/s10741-009-9148-8. PMID 19504345
- [Background] Barghash MH, Lala A, Giustino G, Parikh A, Ullman J, Mitter SS, et al. Use of Remote Dielectric Sensing (ReDS) as Point-of-Care Testing Following Heart Failure Hospitalization and Risk of 30-Day Readmission. J Hear Lung Transplant. 2019;38(4):S140-1
- [Derived] Alvarez-Garcia J, Lala A, Rivas-Lasarte M, De Rueda C, Brunjes D, Lozano-Jimenez S, Garcia-Sebastian C, Mitter S, Remior P, Jimenez-Blanco Bravo M, Del Prado S, Barghash M, Gonzalez-Ferrer E, Ullman J, Cobo M, Segovia-Cubero J, Zamorano JL, Pinney SP, Mancini D. Remote Dielectric Sensing Before and After Discharge in Patients With ADHF: The ReDS-SAFE HF Trial. JACC Heart Fail. 2024 Apr;12(4):695-706. doi: 10.1016/j.jchf.2024.01.002. Epub 2024 Feb 28. PMID 38430084